CLINICAL TRIAL: NCT06864221
Title: Correlation Between Plasma Sphingolipid Metabolites and the Efficacy of Radiotherapy in Hepatocellular Carcinoma
Brief Title: Plasma Sphingolipid Metabolites and Radiotherapy Efficacy in Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-389
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Radiotherapy; Treatment Outcome; Biomarkers; Sphingolipids
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood plasma samples will be collected before, during, and after radiotherapy. The samples will be stored in the institutional biobank at -80°C for lipidomic analysis. After the study, remaining samples will be disposed of according to hospital regulations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiotherapy Responder Group: Participants who show a positive response to radiotherapy, as defined by mRECIST 1.1 criteria. This includes patients with Complete Response (CR) or Partial Response (PR) after radiotherapy. A decline in Alpha-Fetoprotein (AFP) levels may also be observed in some responders, serving as a potential biomarker for treatment efficacy.
- Radiotherapy Non-Responder Group: Participants who do not show a significant response to radiotherapy, as defined by mRECIST 1.1 criteria. This includes patients classified as Stable Disease (SD) or Progressive Disease (PD) after radiotherapy. AFP levels may remain stable or increase in these patients, indicating a lack of significant tumor response to treatment.

SUMMARY:
Plasma contains a variety of metabolites, among which sphingolipids, including ceramide, sphingosine, and sphingosine-1-phosphate, serve as important intracellular second messengers and are involved in various cellular signaling pathways, such as apoptosis. We hypothesize that plasma sphingolipid levels may be associated with the efficacy of radiotherapy for liver cancer. This study will utilize LC-MS/MS technology for qualitative and quantitative analysis of plasma sphingolipids in liver cancer patients undergoing radiotherapy. Clinical data related to patient prognosis will also be collected to investigate the correlation between plasma sphingolipid levels and the therapeutic efficacy of liver cancer radiotherapy. The aim is to establish the clinical diagnostic significance of plasma sphingolipid levels in predicting the efficacy of liver cancer radiotherapy, providing new insights to enhance the effectiveness of radiotherapy in liver cancer treatment.

DETAILED DESCRIPTION:
Liver cancer is one of the most common malignant tumors worldwide, posing a significant challenge to public health. Radiotherapy plays a crucial role in controlling local recurrence and metastasis in hepatocellular carcinoma (HCC) and improving patient survival. Advanced radiotherapy techniques such as Intensity-Modulated Radiation Therapy (IMRT) and Stereotactic Body Radiation Therapy (SBRT) have enhanced tumor dose precision, increasing local control rates while minimizing radiation-induced side effects. However, current methods for assessing radiotherapy efficacy, including CT, MRI, and PET-CT, require extended post-treatment observation periods, delaying clinical decision-making. Additionally, radiotherapy can lead to radiation-induced liver disease (RILD) and other adverse effects such as radiation enteritis and bone marrow suppression. Therefore, identifying early predictive biomarkers for radiotherapy response and toxicity is critical for optimizing treatment strategies.

Sphingolipids, including ceramide (CER), sphingosine (SPH), and sphingosine-1-phosphate (S1P), are essential cellular signaling molecules involved in apoptosis, proliferation, and inflammation. Studies have shown that radiotherapy influences sphingolipid metabolism by altering enzyme activity, thereby affecting the balance of CER, SPH, and S1P-key regulators of tumor cell apoptosis. With advancements in lipidomics, the role of sphingolipid metabolism in radiation sensitivity has become an area of growing interest. Sphingolipid levels have been correlated with radiotherapy sensitivity in various cancers, making them potential prognostic biomarkers and therapeutic targets.

This study is designed as a single-center, prospective observational study with a two-year follow-up period, enrolling 260 primary liver cancer patients receiving radiotherapy. Plasma samples will be collected before, during, and after radiotherapy for qualitative and quantitative analysis of sphingolipid metabolites using liquid chromatography-electrospray ionization-mass spectrometry (LC-ESI-MS). Clinical imaging and laboratory data related to treatment response and adverse events will also be collected. Patients will be classified according to the mRECIST 1.1 criteria into complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) groups for further correlation analysis.

The primary objective is to investigate the relationship between plasma sphingolipid levels and radiotherapy efficacy by analyzing overall survival (OS), objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), disease-free survival (DFS), and time to progression (TTP). The secondary objective is to explore the association between sphingolipid levels and radiation-induced toxicity, including RILD, radiation enteritis, and bone marrow suppression, to assess their potential as predictive biomarkers for treatment-related complications.

Patients will be followed at 1, 2, 6, 12, 18, 24, 36, and 48 months post-radiotherapy. The study does not involve any interventional treatment beyond standard clinical care, and patient management decisions will remain at the discretion of treating physicians. This research aims to provide new insights into the clinical significance of sphingolipid metabolism in predicting radiotherapy outcomes and toxicity in liver cancer, potentially improving personalized radiotherapy strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily signed the informed consent form.
* Aged between 18 and 80 years.
* Clinically diagnosed with primary liver cancer according to the latest treatment guidelines.
* Determined by the treating physician to require radiotherapy.
* Expected survival time of more than 3 months.

Exclusion Criteria:

* Patients who discontinued radiotherapy or did not complete the planned treatment.
* Presence of malignancies from other origins.
* Severe metabolic diseases such as uncontrolled diabetes, significant obesity, or fatty liver disease.
* Uncontrolled comorbidities, such as severe cardiovascular or pulmonary diseases, that may affect treatment or study outcomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients aged 18 to 80 years who have been clinically diagnosed with primary liver cancer according to the latest treatment guidelines. Eligible participants must be determined by their treating physicians to require radiotherapy and have an expected survival time of more than three months. Patients with malignancies of other origins, severe uncontrolled metabolic disorders, or comorbidities that could interfere with treatment outcomes will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From the start of treatment to 12 weeks post-treatment assessment
  Disease Control Rate (DCR) is defined as the proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST). mRECIST is commonly used to evaluate tumor response, especially in the context of hepatocellular carcinoma and other solid tumors. DCR is an important measure to assess the overall effectiveness of the treatment in controlling disease progression.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From treatment initiation to the date of disease progression or death, up to 24 months.
  PFS is defined as the time from the start of treatment to disease progression or death from any cause, whichever occurs first, as assessed by mRECIST. This endpoint measures how long patients remain free from tumor progression.
Overall Survival (OS) | From treatment initiation to death, up to 24 months
  OS is defined as the time from the start of treatment to death from any cause. This endpoint assesses the overall survival benefit of the treatment.
Safety and Tolerability | From the start of treatment until 90 days after the last dose.
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) will be evaluated according to CTCAE (Common Terminology Criteria for Adverse Events) version [specify version]. This endpoint assesses the safety profile of the

CONTACTS AND LOCATIONS:
Overall Officials: Yiyi Li, PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Due to ethical and privacy concerns, the individual participant data (IPD) will not be shared. All data will be anonymized and stored securely to protect participants' privacy, as per institutional guidelines. Sharing IPD may pose a risk of re-identification or misuse of personal information, which could potentially violate the confidentiality agreement with the participants. Therefore, the data will remain confidential and only be used for the specific purposes outlined in the study protocol.

REFERENCES:
- [Result] Deng X, Yin X, Allan R, Lu DD, Maurer CW, Haimovitz-Friedman A, Fuks Z, Shaham S, Kolesnick R. Ceramide biogenesis is required for radiation-induced apoptosis in the germ line of C. elegans. Science. 2008 Oct 3;322(5898):110-5. doi: 10.1126/science.1158111. PMID 18832646
- [Result] Kumar A, Oskouian B, Fyrst H, Zhang M, Paris F, Saba JD. S1P lyase regulates DNA damage responses through a novel sphingolipid feedback mechanism. Cell Death Dis. 2011 Feb 10;2(2):e119. doi: 10.1038/cddis.2011.3. PMID 21368890
- [Result] Taha TA, Osta W, Kozhaya L, Bielawski J, Johnson KR, Gillanders WE, Dbaibo GS, Hannun YA, Obeid LM. Down-regulation of sphingosine kinase-1 by DNA damage: dependence on proteases and p53. J Biol Chem. 2004 May 7;279(19):20546-54. doi: 10.1074/jbc.M401259200. Epub 2004 Feb 26. PMID 14988393
- [Result] Aureli M, Bassi R, Prinetti A, Chiricozzi E, Pappalardi B, Chigorno V, Di Muzio N, Loberto N, Sonnino S. Ionizing radiations increase the activity of the cell surface glycohydrolases and the plasma membrane ceramide content. Glycoconj J. 2012 Dec;29(8-9):585-97. doi: 10.1007/s10719-012-9385-2. Epub 2012 May 17. PMID 22592846
- [Result] Cheng JC, Bai A, Beckham TH, Marrison ST, Yount CL, Young K, Lu P, Bartlett AM, Wu BX, Keane BJ, Armeson KE, Marshall DT, Keane TE, Smith MT, Jones EE, Drake RR Jr, Bielawska A, Norris JS, Liu X. Radiation-induced acid ceramidase confers prostate cancer resistance and tumor relapse. J Clin Invest. 2013 Oct;123(10):4344-58. doi: 10.1172/JCI64791. Epub 2013 Sep 16. PMID 24091326
- [Result] Garcia-Barros M, Paris F, Cordon-Cardo C, Lyden D, Rafii S, Haimovitz-Friedman A, Fuks Z, Kolesnick R. Tumor response to radiotherapy regulated by endothelial cell apoptosis. Science. 2003 May 16;300(5622):1155-9. doi: 10.1126/science.1082504. PMID 12750523
- [Result] Liao WC, Haimovitz-Friedman A, Persaud RS, McLoughlin M, Ehleiter D, Zhang N, Gatei M, Lavin M, Kolesnick R, Fuks Z. Ataxia telangiectasia-mutated gene product inhibits DNA damage-induced apoptosis via ceramide synthase. J Biol Chem. 1999 Jun 18;274(25):17908-17. doi: 10.1074/jbc.274.25.17908. PMID 10364237
- [Result] Gomez-Larrauri A, Presa N, Dominguez-Herrera A, Ouro A, Trueba M, Gomez-Munoz A. Role of bioactive sphingolipids in physiology and pathology. Essays Biochem. 2020 Sep 23;64(3):579-589. doi: 10.1042/EBC20190091. PMID 32579188
- [Result] Benson R, Madan R, Kilambi R, Chander S. Radiation induced liver disease: A clinical update. J Egypt Natl Canc Inst. 2016 Mar;28(1):7-11. doi: 10.1016/j.jnci.2015.08.001. Epub 2015 Aug 20. PMID 26300327
- [Result] Wen N, Cai Y, Li F, Ye H, Tang W, Song P, Cheng N. The clinical management of hepatocellular carcinoma worldwide: A concise review and comparison of current guidelines: 2022 update. Biosci Trends. 2022 Mar 11;16(1):20-30. doi: 10.5582/bst.2022.01061. Epub 2022 Feb 24. PMID 35197399
- [Result] Vogel A, Meyer T, Sapisochin G, Salem R, Saborowski A. Hepatocellular carcinoma. Lancet. 2022 Oct 15;400(10360):1345-1362. doi: 10.1016/S0140-6736(22)01200-4. Epub 2022 Sep 6. PMID 36084663